CLINICAL TRIAL: NCT01554553
Title: A Prospective Randomized Clinical Trial Comparing Patients Who Have Had Longitudinal Sleeve Gastrectomy With Posterior Crural Repair Versus Without Posterior Crural Repair
Brief Title: Longitudinal Sleeve Gastrectomy Study Comparing Posterior Crural Repair Versus No Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Brad Snyder, MD - Principal Investigator, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HSC-MS-11-0605
Record Dates: First submitted 2012-02-24; First posted 2012-03-15 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Obesity
Keywords: Sleeve gastrectomy; Posterior crural repair
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Posterior crural repair (Experimental)
  Interventions: Procedure: Posterior crural repair
- No posteriorcrural repair (No Intervention)

INTERVENTIONS:
Procedure: Posterior crural repair — All patients receive gastrectomy, however patients randomized to the experimental arm will also receive posterior crural repair to determine if this will reduce GERD post sleeve gastrectomy.
  Other Names: gastric sleeve with crural repair
  Arms: Posterior crural repair

SUMMARY:
The purpose of this study is to evaluate the superiority of posterior crural repair during sleeve gastrectomy over no repair in decreasing the incidence of symptomatic and clinical reflux disease.

DETAILED DESCRIPTION:
Longitudinal Sleeve gastrectomy is a type of Bariatric surgery where the stomach is divided vertically, reducing it to about 25% of its original size. Obesity itself is an independent risk factor for Gastroesophageal reflux disease (GERD); however it has been observed in the bariatric surgical community that many Longitudinal Sleeve Gastrectomy (LSG) patients are complaining of persisted GERD symptoms after LSG surgery. The incidence of GERD in these patients have been reported to be as high as 26%. GERD is an uncomfortable and dangerous disease, and if remains unchecked, it can cause ulcer disease, esophagitis, and even esophageal cancer. Because of this, bariatric surgeons want to reduce incidence of GERD after LSG, which led to multiple additions to the LSG procedures, which are currently being examined, namely, combined fundoplication with the sleeve, banded sleeve and a combined hiatal repair with SG. However, there have been no randomized comparative clinical trials to evaluate GERD as an endpoint after LSG.

Of all the possible solutions to treat increased reflux after LSG, mentioned previously, repairing the hiatus at the time of surgery makes the most sense physiologically. LSG dissection requires the obliteration of the left phrenoesophageal ligaments that hold the GE junction in place. This essentially creates a weakness in the hiatus that can lead to hiatal hernia and subsequent reflux disease. Crural repair at the time of surgery strengthens the GE junction and reduces the possibility of hiatal hernia formation. Closing the crus around the esophagus may prevent the sleeve from herniating into the chest and reduces the occurrence of reflux by repositioning the GE junction into it0s normal location in the abdomen.

ELIGIBILITY:
INCLUSION CRITERIA:

* The subject is between the ages of 21 and 65
* The subject is able to provide informed consent
* The subject is able and willing to comply with the study protocol
* Patients are will to refrain from the use of specified antacid medications such as PPIs (e.g. Nexium, Prilosec, Omeprazole, etc) or H2 blockes (e.g. Pepcid, Zantac, etc)
* The subjects meets the requirement for bariatric surgery as defined by the 1991 NIH consensus on bariatric surgery
* BMI ≥40 or BMI = 35-39 with one or more obesity-related comorbidities.
* Patients should have attempted, and failed, several structured methods of weight loss The subject is approved to have a sleeve gastrectomy

EXCLUSION CRITERIA:

* The subject is not able to provide informed consent
* The subject is not willing to comply with the study protocol
* The subject has had previous foregut (stomach) surgery
* The subject has evidence of a gastric tumor, ulcer, or other abnormalities at the time of EGD that would preclude them from having a sleeve gastrectomy
* Severe esophagitis or Barrett's esophagus will exclude them from the study
* The surgeon concludes that the patient is not a candidate for sleeve gastrectomy based on his clinical judgment

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Change in GERD / GSRS Quality of Life Questionnaire | 1 questionnaire pre-operatively, and then every 3 months for the 1st year, every 6 months until the third year, and every 12 months until 6 years.
  The primary outcome of the study will be the patients' self-assessment of their reflux symptoms as reported with the GSRS quality of life questionnaire that was specifically designed to be used as an outcome measure in clinical trials of intervention in GERD. The final primary outcome will be measured every year to assess allieviation or change of reflux sysmtpms over time and to ensure there is no reoccurence of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Brad Snyder, MD, Principal Investigator — UT Medical School at Houston, Dept. of Surgery
Locations (1):
- Minimally Invasive Surgeons of Texas (MIST), Bariatric Clinic, Houston, Texas, United States